CLINICAL TRIAL: NCT06165744
Title: Next Generation Cataract and Vitreoretinal Surgery Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTV678-E001
Record Dates: First submitted 2023-12-04; First posted 2023-12-11 (Actual); Results first posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Vitreoretinal Disease With or Without Cataracts
Keywords: Vitreoretinal surgery; Vitreoretinal with cataract surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- UNITY VCS (Experimental): Posterior segment surgery in the operating room with or without simultaneous cataract surgery performed with UNITY VCS
  Interventions: Device: UNITY Vitreoretinal Cataract System; Procedure: Posterior segment surgery in the operating room with or without simultaneous cataract surgery

INTERVENTIONS:
Device: UNITY Vitreoretinal Cataract System — UNITY Vitreoretinal Cataract System (VCS) with console, remote control, foot controller, UNITY TOTAL PLUS Combined Procedure Pak, and additional devices as needed to complete surgery
  Other Names: UNITY VCS
Procedure: Posterior segment surgery in the operating room with or without simultaneous cataract surgery — Posterior segment surgery involves removal of the vitreous (i.e., vitrectomy) followed by additional interventions as needed. Cataract surgery involves removal of the crystalline lens (which is often cloudy).

SUMMARY:
The purpose of this study is to obtain device-specific safety and performance clinical data to support marketability in Europe and to collect formal user feedback.

DETAILED DESCRIPTION:
Subjects will attend a screening visit (Day -30 to Day 0), a surgery visit (Day 0), and 4 post-surgical visits (Day 1, Week 1, Month 1, Month 3) for an overall individual duration of approximately 4 months. One eye (study eye) will be treated. This study will be conducted in Australia.

ELIGIBILITY:
Key Inclusion Criteria:

* Requires posterior segment surgery in the operating room with or without simultaneous cataract surgery;
* Clear media except for cataract and vitreous hemorrhage;
* In simultaneous cataract and vitreoretinal surgery, eligible to undergo primary hydrophobic acrylic intraocular lens (IOL) implantation into the capsular bag;
* Other protocol-defined inclusion criteria may apply.

Key Exclusion Criteria:

* Previous vitrectomy in the operative eye aside from those requiring silicone oil removal;
* Neovascular or uncontrolled glaucoma;
* Planned glaucoma or postoperative surgeries during study aside from silicone oil removal;
* Inadequate pupil dilation (less than 6 millimeters);
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2024-02-27 (Actual); Primary Completion 2024-05-23 (Actual); Study Completion 2024-08-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sr. Clinical Operations Lead, Surgical, Study Director — Alcon Research, LLC
Locations (5):
- Australia (5):
  - NSW Retina Pty Ltd, Hurstville, New South Wales
  - Southwest Retina, Liverpool, New South Wales
  - Sydney Retina Clinic & Day Surgery, Sydney, New South Wales
  - Adelaide Eye & Retina Centre, Adelaide, South Australia
  - Pennington Eye Clinic, North Adelaide, South Australia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 5 investigative sites located in Australia.
Pre-assignment Details: Of the 120 participants enrolled in the study, 2 were exited as screen failures, resulting in 118 participants treated. This reporting group includes all treated participants.
Units Other Than Participants: eyes
Period: Overall Study
Arm/Group | UNITY VCS
Started | 118; 118 eyes
Completed | 117; 117 eyes
Not Completed | 1; 1 eyes
Not completed — Non device-related adverse event | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: All eyes with attempted use of the UNITY VCS (successful or aborted after contact with the eye).
Arm/Group | UNITY VCS
Number analyzed (Participants) | 118
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.5 (13.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52
  Male | 66
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 115
  Unknown or Not Reported | 1
Race/Ethnicity, Customized [Number; unit: participants]
  White | 91
  Black or African American | 0
  American Indian or Alaska Native | 0
  Asian | 16
  Native Hawaiian or Other Pacific Islander | 5
  Other | 6
Region of Enrollment [Number; unit: participants]
  Australia | 118

OUTCOME MEASURES:

1. Primary Outcome: Percent of 'Yes' Responses to the Binary Question: "Did UNITY VCS Using Vitreoretinal or Combined Surgical Functionality Perform Per the Intended Use as Defined in Protocol Section 5.1?"
Description: As recorded by the surgeon on a user questionnaire based on Day 0 surgery experience. From Protocol Section 5.1, the intended use for UNITY VCS is to facilitate the management of fluid and gases, as well as removal, grasping, cutting, illumination, and coagulation of ocular materials during ocular surgery. One eye (study eye) contributed data to the analysis. No hypothesis testing was pre-specified for this endpoint.
Time Frame: Day 0
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of responses
Units Other Than Participants: eyes
Arm/Group | UNITY VCS
Number analyzed (Participants) | 117
Number analyzed (eyes) | 117
percentage of responses | 100 [96.9 to 100]

2. Secondary Outcome: Mean Total Time in Eye
Description: The time from first entry into eye/first trocar in to incision closure/last trocar out was measured using a stopwatch and recorded in minutes. One eye (study eye) contributed data to the analysis. No hypothesis testing was pre-specified for this endpoint.
Time Frame: Day 0 operative, up to surgery completion
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: minutes
Units Other Than Participants: eyes
Arm/Group | UNITY VCS
Number analyzed (Participants) | 117
Number analyzed (eyes) | 117
minutes | 22.788 (11.5663)

3. Secondary Outcome: Percent of 'Yes' Responses to the Binary Question, "Was Anatomical Success Achieved for Intended Treatment?"
Description: As reported by the examiner at the Month 3 visit. Intended treatment included macular hole closure, retinal attachment, etc. as applicable for the patient's condition. One eye (study eye) contributed data to the analysis. No hypothesis testing was pre-specified for this endpoint.
Time Frame: Month 3 Postoperative
Population: Full Analysis Set with data at Month 3 visit
Measure: Number (95% Confidence Interval); unit: percentage of responses
Units Other Than Participants: eye
Arm/Group | UNITY VCS
Number analyzed (Participants) | 116
Number analyzed (eye) | 116
percentage of responses | 96.6 [91.4 to 99.1]

4. Secondary Outcome: Mean Change in Monocular Best Corrected Distance Visual Acuity (BCDVA) From Preoperative to Month 3
Description: Visual acuity was assessed with refractive correction in place using a Snellen visual acuity chart. Results were converted to decimal VA, where 2.00 decimal equates to 20/16 Snellen (better than normal distance eyesight), 1.00 decimal equates to 20/20 Snellen (normal distance eyesight), and 0.1 decimal equates to 6/600 Snellen (worse than normal distance eyesight). A positive change value indicates an improvement. One eye (study eye) contributed data to the analysis. No hypothesis testing was pre-specified for this endpoint.
Time Frame: Preoperative (Day -30 to 0), Month 3 Postoperative
Population: Full Analysis Set with numerical Snellen values at both Preoperative and Month 3 visits
Measure: Mean (Standard Deviation); unit: decimal
Units Other Than Participants: eyes
Arm/Group | UNITY VCS
Number analyzed (Participants) | 99
Number analyzed (eyes) | 99
decimal | 0.186 (0.2410)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from time of consent to study exit, up to approximately 4 months
Description: AEs were obtained through solicited and spontaneous comments from the subjects and through observations by the investigator. This analysis population includes all subjects/eyes with attempted use of the UNITY VCS (successful or aborted after contact with the eye). The Other (Not Including Serious) Adverse Event table reports only the AEs that occurred above a 5% threshold in one or more reporting groups.
Groups:
- Pretreatment: AEs in this group occurred prior to treatment with UNITY VCS
- UNITY VCS Ocular - Study Eye: AEs in this group occurred after attempted treatment with with UNITY VCS and include ocular events in the study eye. "At Risk" population is reported in units of eyes.
- UNITY VCS Systemic: AEs in this group occurred after attempted treatment with UNITY VCS and include overall systemic events as well as ocular events in the non-study eye. "At Risk" population is reported in units of subjects.
Arm/Group | Pretreatment | UNITY VCS Ocular - Study Eye | UNITY VCS Systemic
All-Cause Mortality (participants affected / at risk) | 0/118 | 0/118 | 0/118
Serious Adverse Events (participants affected / at risk) | 1/118 | 38/118 | 6/118
Other Adverse Events (participants affected / at risk) | 0/118 | 21/118 | 1/118
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pretreatment (N=118) | UNITY VCS Ocular - Study Eye (N=118) | UNITY VCS Systemic (N=118)
Cystoid macular oedema (Eye disorders) | 0 (0) | 3 (3) | 0 (0)
Diabetic retinal oedema (Eye disorders) | 0 (0) | 1 (1) | 2 (2)
Epiretinal membrane (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotony of eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Iris disorder (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Macular hole (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Macular oedema (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Pupillary block (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 8 (10) | 0 (0)
Retinal disorder (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Retinal haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 2 (2)
Retinal oedema (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Retinal tear (Eye disorders) | 0 (0) | 11 (11) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 8 (8) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Intraocular pressure increased (Investigations) | 0 (0) | 5 (5) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Haemorrhage urinary tract (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Intra-ocular injection (Surgical and medical procedures) | 0 (0) | 6 (9) | 0 (0)
Iridotomy (Surgical and medical procedures) | 0 (0) | 1 (2) | 0 (0)
Retinal operation (Surgical and medical procedures) | 0 (0) | 9 (10) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pretreatment (N=118) | UNITY VCS Ocular - Study Eye (N=118) | UNITY VCS Systemic (N=118)
Cataract (Eye disorders) | 0 (0) | 7 (7) | 0 (0)
Intraocular pressure increased (Investigations) | 0 (0) | 15 (15) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2024-02-04): https://cdn.clinicaltrials.gov/large-docs/44/NCT06165744/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-06): https://cdn.clinicaltrials.gov/large-docs/44/NCT06165744/SAP_001.pdf